CLINICAL TRIAL: NCT05256082
Title: Impact of Face Masks on the Six Minute Walking Distance in Pulmonary Hypertension Patients During the COVID-19 Pandemic: A Prospective, Randomized Cross-over Study
Brief Title: Impact of Face Masks on 6MWD in Patients With Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Max Wissmueller, Dr. med. Max Wissmueller, University Hospital of Cologne
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020_01; UoC Ethics 20-1581-1 (Other: University Hospital of Cologne)
Record Dates: First submitted 2020-11-04; First posted 2022-02-25 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; exercise capacity; six minute walking distance; face mask; COVID-19
MeSH Terms: conditions — Hypertension, Pulmonary; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- with mask (FFP2 mask or surgical mask) (Active Comparator): Patient is Walking with mouth/nose-mask for 6 Minutes.
  Interventions: Diagnostic Test: six-minutes-walking test
- without mask (Placebo Comparator): Patient is Walking without mouth/nose-mask for 6 Minutes.
  Interventions: Diagnostic Test: six-minutes-walking test

INTERVENTIONS:
Diagnostic Test: six-minutes-walking test — Patients conducting a six-minutes-walking test

SUMMARY:
Pulmonary hypertension (PH) is classified according to the Nice Classification into different etiologies, including pulmonary arterial hypertension (PAH), a disease of the pulmonary arteriolar vasculature (Class I), and forms of pulmonary hypertension associated with left heart disease (Class II), lung disease (Class III), pulmonary artery obstructions including chronic pulmonary embolism (Class IV) or other less common causes (Class V). Patients with PH are at risk in the current COVID 19 pandemic.

The course of the disease and the prognosis of the patients are assessed on the basis of various parameters and therapy is adapted accordingly. In addition to clinical, echocardiographic and laboratory examinations, cardiopulmonary performance tests such as the 6-minute walking distance (6MWD) are of particular significance. According to the ESC/ERS guidelines for PH and the recommendations of the Cologne Consensus Conference, exercise performance is a central criterion for prognostication and treatment decisions.

During the COVID-19 pandemic, hospitals require the constant use of face masks for patients, in most cases also during the 6 minute walking test. We suspect a performance-reducing effect of face masks, thus impacting the results of the 6MWD. A systematic error in the assessment of cardiopulmonary performance should be revealed by comparing the results of the 6MWD with and without mask (particularly surgical mask and FFP2 mask).

DETAILED DESCRIPTION:
Monocentric, prospective, randomized cross-over study in approximately 120 patients with PH (n=60 for surgical face mask versus no mask; n=60 for FFP2 mask vs. no mask) to evaluate the impact of face masks on 6MWD, Borg dyspnea score, and O2 saturation pre- versus post exercise. Patients are randomized to perform the test with vs. without mask first, and then cross over to the respective other condition.

The primary endpoint is the intra-individual difference in 6MWD with and without mask (analyzed for the whole study group, and for surgical mask and FFP2 mask seperately). Secondary endpoints include differences in Borg score, and O2 saturation.

ELIGIBILITY:
Inclusion Criteria:

* Regular 6MWD in the last 24 months, at least 1 test per 24 months
* Pulmonary (arterial) hypertension according to the Nice Classification Type I-V
* NYHA-WHO/FC I - III
* Lung function test performed within 6 months
* Age ≥18 years
* Severity of symptoms and specific therapy stable during the last 4 weeks
* General ability to participate in the study
* Ability to give consent

Exclusion Criteria:

* Contact allergy to face mask materials
* Significant peripheral arterial occlusive disease (Fontaine ≥ IIb)
* Muscular or orthopedic diseases of the lower extremities that contribute to reduced resilience
* Relevant coronary heart disease (angina pectoris ≥ CCS II or positive stress test, myocardial infarction or bypass surgery within the last 3 months)
* inability to perform the 6-minute walk test (mental, physical) or lack of ability to provide essential information (questionnaire, Borg level)
* Uncontrolled high blood pressure (≥140/90 mmHg or ≥160/100 mmHg with 3 antihypertensive drugs) or resting heart rate ≥ 100 b.p.m.)
* Fresh fractures / broken bones (within the last 3 months)
* Not able to give consent Insufficient ability to walk (NYHA IV, immobility, other ailments)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Intra-individual difference in six-minute-walking-distance (6MWD) with versus without face mask | one day while follow-up visit in PAH-center
  Patients repeat a walking-test, conducting 2 walks on one day while a Follow-Up-visit. Change in six-minutes-walking-distance will be measured intra-individually. Patients are walking without mask (control) and wearing a mask (intervention). Minimum 1 hour of rest in between control and intervention. A cross-over design is performed with randomization, if mask will be used in the first six-minutes-walking.

SECONDARY OUTCOMES:
PAH-specific Quality of life Baseline | while follow-up 1 day visit in PAH-center
  PAH-specific Quality of life assessed by PAH-Sympact (Pulmonary Arterial Hypertension-Symptoms and Impact Questionnaire)
Depression Baseline | while follow-up 1 day visit in PAH-center
  Depression assessed by PHQ9 (Patient Health Questionnaire, 1-27 points with higher depression-severity with higher total points)
Anxiety Baseline | while follow-up 1 day visit in PAH-center
  Anxiety assessed by GAD7 (Generalized Anxiety Disorder Scale 7; 0-21 points with higher Anxiety-Symptoms with higher total points)
Intra-individual difference in pSO2 performing a six-minutes-walking-test (6MWT) with face mask | one day while follow-up-visit in PAH-center
  Patients repeat a walking-test, conducting 2 walks on one day while a Follow-Up-visit. Change in pSO2 while the six-minutes-walking-test will be measured intra-individually. Patients are walking without mask (control) and wearing a mask (intervention). Minimum 1 hour of rest in between control and intervention. A cross-over design is performed with randomization, if mask will be used in the first six-minutes-walking.
  The pSO2 is continuously documented while patients perform the walking test and while the first 3 Minutes of rest after walking.
Intra-individual difference in Borg dyspnea score after a six-minutes-walking-test (6MWT) with versus without face mask | one day while follow-up-visit in PAH-center
  Patients repeat a walking-test, conducting 2 walks on one day while a Follow-Up-visit. Dyspnea is assessed by Borg dyspnea score (Borg dyspnea score; 0-10 points with increasing dyspnea-severity with higher total points)

CONTACTS AND LOCATIONS:
Overall Officials: Max VJ Wissmueller, MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tschope C, Birner C, Bohm M, Bruder O, Frantz S, Luchner A, Maier L, Stork S, Kherad B, Laufs U. Heart failure with preserved ejection fraction: current management and future strategies : Expert opinion on the behalf of the Nucleus of the "Heart Failure Working Group" of the German Society of Cardiology (DKG). Clin Res Cardiol. 2018 Jan;107(1):1-19. doi: 10.1007/s00392-017-1170-6. Epub 2017 Oct 10. PMID 29018938
- [Background] Eikenberry SE, Mancuso M, Iboi E, Phan T, Eikenberry K, Kuang Y, Kostelich E, Gumel AB. To mask or not to mask: Modeling the potential for face mask use by the general public to curtail the COVID-19 pandemic. Infect Dis Model. 2020 Apr 21;5:293-308. doi: 10.1016/j.idm.2020.04.001. eCollection 2020. PMID 32355904
- [Background] Greenhalgh T, Schmid MB, Czypionka T, Bassler D, Gruer L. Face masks for the public during the covid-19 crisis. BMJ. 2020 Apr 9;369:m1435. doi: 10.1136/bmj.m1435. No abstract available. PMID 32273267
- [Background] Liang M, Gao L, Cheng C, Zhou Q, Uy JP, Heiner K, Sun C. Efficacy of face mask in preventing respiratory virus transmission: A systematic review and meta-analysis. Travel Med Infect Dis. 2020 Jul-Aug;36:101751. doi: 10.1016/j.tmaid.2020.101751. Epub 2020 May 28. PMID 32473312
- [Background] Lyu W, Wehby GL. Community Use Of Face Masks And COVID-19: Evidence From A Natural Experiment Of State Mandates In The US. Health Aff (Millwood). 2020 Aug;39(8):1419-1425. doi: 10.1377/hlthaff.2020.00818. Epub 2020 Jun 16. PMID 32543923
- [Background] Worby CJ, Chang HH. Face mask use in the general population and optimal resource allocation during the COVID-19 pandemic. Nat Commun. 2020 Aug 13;11(1):4049. doi: 10.1038/s41467-020-17922-x. PMID 32792562
- [Background] Roberge RJ, Kim JH, Benson SM. Absence of consequential changes in physiological, thermal and subjective responses from wearing a surgical mask. Respir Physiol Neurobiol. 2012 Apr 15;181(1):29-35. doi: 10.1016/j.resp.2012.01.010. Epub 2012 Feb 2. PMID 22326638
- [Background] Roberge RJ, Coca A, Williams WJ, Palmiero AJ, Powell JB. Surgical mask placement over N95 filtering facepiece respirators: physiological effects on healthcare workers. Respirology. 2010 Apr;15(3):516-21. doi: 10.1111/j.1440-1843.2010.01713.x. Epub 2010 Mar 11. PMID 20337987
- [Background] Li R, Pei S, Chen B, Song Y, Zhang T, Yang W, Shaman J. Substantial undocumented infection facilitates the rapid dissemination of novel coronavirus (SARS-CoV-2). Science. 2020 May 1;368(6490):489-493. doi: 10.1126/science.abb3221. Epub 2020 Mar 16. PMID 32179701
- [Background] Fikenzer S, Laufs U. Response to Letter to the editors referring to Fikenzer, S., Uhe, T., Lavall, D., Rudolph, U., Falz, R., Busse, M., Hepp, P., & Laufs, U. (2020). Effects of surgical and FFP2/N95 face masks on cardiopulmonary exercise capacity. Clinical research in cardiology: official journal of the German Cardiac Society, 1-9. Advance online publication. https://doi.org/10.1007/s00392-020-01704-y. Clin Res Cardiol. 2020 Dec;109(12):1600. doi: 10.1007/s00392-020-01736-4. Epub 2020 Sep 23. No abstract available. PMID 32989474
- [Derived] Wissmuller M, Wartner V, Hohmann C, Adler J, Kramer T, Hellmich M, Gerhardt F, Baldus S, Rosenkranz S. Impact of face masks on the 6-minute walk distance in pulmonary hypertension patients during the COVID-19 pandemic: a prospective, randomised cross-over study. Eur Respir J. 2023 Oct 26;62(4):2201454. doi: 10.1183/13993003.01454-2022. Print 2023 Oct. PMID 37827573